CLINICAL TRIAL: NCT06250426
Title: REFRESH Study: Therapeutic Effect of a Cooling Sensation Flavor in Pre-thickened ONS Products on the Swallow Response in Post-stroke Patients With Oropharyngeal Dysphagia
Brief Title: Effect of a Cooling Sensation Flavor on the Swallow Response in Post-stroke Patients With Oropharyngeal Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Principal Investigator, Pere Clave, Principal Investigator, Hospital de Mataró
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Refresh
Record Dates: First submitted 2023-07-06; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Oropharyngeal Dysphagia; Stroke; Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, interventional and, open-label clinical study. The study includes 2 groups: 1) n=25: 1st visit: stimulation with Control, 2nd visit: stimulation with CS; and 2) n=25: 1st visit: stimulation with CS, 2nd visit: stimulation with Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Pre-thickened oral nutritional supplement with a cooling sensation flavour
  Interventions: Dietary Supplement: Pre-thickened oral nutritional supplement with a cooling sensation flavour
- Control (Placebo Comparator): Pre-thickened oral nutritional supplement without a cooling sensation flavour
  Interventions: Dietary Supplement: Pre-thickened oral nutritional supplement without a cooling sensation flavour

INTERVENTIONS:
Dietary Supplement: Pre-thickened oral nutritional supplement with a cooling sensation flavour — Pre-thickened oral nutritional supplement (ONS) drink with cooling sensation flavour
  Arms: Active
Dietary Supplement: Pre-thickened oral nutritional supplement without a cooling sensation flavour — Pre-thickened oral nutritional supplement (ONS) drink without cooling sensation flavour
  Arms: Control

SUMMARY:
Current oropharyngeal dysphagia (OD) treatment in older patients is based on compensatory strategies (fluid thickening and texture modified diets) that improve swallow safety but do not improve the swallowing function. One of these strategies is thickening products, which are used to reduce pharyngeal bolus velocity by increasing viscosity of fluids. There are several studies demonstrating the therapeutic effect of thickeners in reducing the prevalence of penetrations and aspirations, and their use has been correlated with reduced prevalence of respiratory infections, aspiration pneumonia and hospital readmissions.

In recent years, new neurorehabilitation treatment strategies for OD have been developed such as peripheral (electrical or chemical stimulation) or central stimulation (transcranial direct current stimulation or repetitive transcranial magnetic stimulation).

The investigators suggest that new generation treatments for OD have to combine thickened fluids and about peripheral stimulation using transient receptor potential (TRP) channels agonists. The aim of this study is to evaluate the therapeutic effect of a cooling sensation (CS) flavor in a pre-thickened oral nutritional supplement (ONS) drink on the biomechanical mechanism of the swallow response in chronic post-stroke patients with OD.

The investigators designed a randomized, crossover, interventional and open-label clinical study. The study includes 2 groups: 1) n=25: 1st visit: stimulation with Control, 2nd visit: stimulation with CS; and 2) n=25: 1st visit: stimulation with CS, 2nd visit: stimulation with Control. Each patient will attend a total of 2 visits, with a washing period of at least 7 days between visits. The procedures to be performed during each visit are: clinical assessment of swallowing with V-VST, spontaneous swallowing frequency measurement using electromyography, and collection of a sample of saliva using a Salivette®.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Patients with chronic OD as a consequence of stroke (more than 3 month since stroke diagnostic)
* Patients with impaired safety and/or efficacy of swallow (V-VST)
* Patients that can swallow safely the investigation and control product according to the viscosity of the product and the results of the V-VST
* Patients able to follow the protocol and give informed consent

Exclusion Criteria:

* Pregnancy
* Life expectancy <3 months or palliative care
* OD diagnosis prior to stroke
* Dementia (GDS 4 or higher)
* Allergy to the investigation and/or control product or to any of its components
* Participation in another interventional study in the month prior to inclusion
* Current users of a pre-thickened ONS drink with cooling sensation flavor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Pre visit 1 Spontaneous swallowing frequency (SSF) | Pre intervention in visit 1 (baseline)
  SSF will be measured with surface neck electromyography (sEMG) and accelerometry for 10min, in which the patient will be asked to breathe normally and to remain calm and quiet. sEMG electrodes will be placed over the digastric-mylohyoid complex and an omnidirectional accelerometer over the cricothyroid cartilage to assess the number of swallows per minute.
Pre visit 1 EMG metrics | Pre intervention in visit 1 (baseline)
  EMG metrics (amplitude (Volts), latency (seconds), duration (seconds) and area under the curve (volts·second)) of the recordings using the AcqKnowledge 4.4 software (BIOPAC Systems, USA) will be analyzed and combined to describe the electromyographic response of the suprahyoid muscles.
Post visit 1 Spontaneous swallowing frequency (SSF) | Post intervention in visit 1 (baseline)
  SSF will be measured with surface neck electromyography (sEMG) and accelerometry for 10min, in which the patient will be asked to breathe normally and to remain calm and quiet. sEMG electrodes will be placed over the digastric-mylohyoid complex and an omnidirectional accelerometer over the cricothyroid cartilage to assess the number of swallows per minute.
Post visit 1 EMG metrics | Post intervention in visit 1 (baseline)
  EMG metrics (amplitude (Volts), latency (seconds), duration (seconds) and area under the curve (volts·second)) of the recordings using the AcqKnowledge 4.4 software (BIOPAC Systems, USA) will be analyzed and combined to describe the electromyographic response of the suprahyoid muscles.
Pre visit 2 Spontaneous swallowing frequency (SSF) | Pre intervention visit 2 (1 week after)
  SSF will be measured with surface neck electromyography (sEMG) and accelerometry for 10min, in which the patient will be asked to breathe normally and to remain calm and quiet. sEMG electrodes will be placed over the digastric-mylohyoid complex and an omnidirectional accelerometer over the cricothyroid cartilage to assess the number of swallows per minute.
Pre visit 2 EMG metrics | Pre intervention visit 2 (1 week after)
  EMG metrics (amplitude (Volts), latency (seconds), duration (seconds) and area under the curve (volts·second)) of the recordings using the AcqKnowledge 4.4 software (BIOPAC Systems, USA) will be analyzed and combined to describe the electromyographic response of the suprahyoid muscles.
Post visit 2 Spontaneous swallowing frequency (SSF) | Post intervention visit 2 (1 week after)
  SSF will be measured with surface neck electromyography (sEMG) and accelerometry for 10min, in which the patient will be asked to breathe normally and to remain calm and quiet. sEMG electrodes will be placed over the digastric-mylohyoid complex and an omnidirectional accelerometer over the cricothyroid cartilage to assess the number of swallows per minute.
Post visit 2 EMG metrics | Post intervention visit 2 (1 week after)
  EMG metrics (amplitude (Volts), latency (seconds), duration (seconds) and area under the curve (volts·second)) of the recordings using the AcqKnowledge 4.4 software (BIOPAC Systems, USA) will be analyzed and combined to describe the electromyographic response of the suprahyoid muscles.

SECONDARY OUTCOMES:
Volume-viscosity swallowing test (V-VST) | Pre and Post treatment in visit 1 (baseline) and visit 2 (1 week after)
  The V-VST is an effort test in which boluses of increasing volume and viscosity are administered to check for clinical signs of impaired efficacy and safety in each swallow. V-VST is designed to protect patients from aspiration by starting with 250 mPa•s viscosity and increasing volumes from 5 ml, to 10 ml and 20 ml boluses. When patients have completed the 250 mPa•s series without major symptoms of aspiration, a less safe liquid viscosity series will be assessed. Finally, a safer 800 mPa•s viscosity series will be assessed in the same way. If the patient presents signs of impaired safety at 250 mPa•s viscosity, the series will be interrupted, the <50 mPa•s viscosity series will be omitted, and a safer 800 mPa•s viscosity series will be assessed. If the patient presents signs of impaired safety at <50 mPa•s viscosity, the liquid series will be interrupted, and the 800 mPa•s series will be assessed.
Concentration of salivary neuropeptides | Pre and Post treatment in visit 1 (baseline) and visit 2 (1 week after)
  Saliva samples will be collected using the Salivette® technique, by putting a swab under the tongue for 5 min. Samples will be stored at -80ºC until their analysis. The concentration of salivary neuropeptides substance P (SP) and calcitonin gene-related peptide (CGRP) will be determined by using 2 specific commercial Enzyme-Linked ImmunoSorbent Assay (ELISA) kits: Substance P Parameter Assay Kit (R&D systems, USA) and CGRP (Human) ELISA kit (Abnova, Taiwan).

OTHER OUTCOMES:
Characterization of the rheological properties of the study products | Previous to the start of the clinical study
  Determination of the viscosity in mPa•s at 50s-1 and the effect of the shear rate (viscosity at 50s-1 and at 300s-1) and alpha-amylase will be determine for both products.
  The rheological data will ensure the safety of the patients with OD during the study procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No